CLINICAL TRIAL: NCT06884631
Title: Metabolic Exercise Test Data Combined with Cardiac and Kidney Indexes (MECKI) Score Evolution: Study of Cardiovascular Risk in Patients with Heart Failure
Brief Title: Metabolic Exercise Test Data Combined with Cardiac and Kidney Indexes (MECKI) Score Evolution: Identification of Cardiovascular Risk in Patients with Heart Failure
Acronym: MECKI
Status: Recruiting | Type: Observational
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Santo Spirito Hospital, Italy (Other); Fondazione Toscana Gabriele Monasterio (Other); Spedali Civili, University of Brescia, Italy (Unknown); Monaldi Hospital (Other); Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI) (Unknown); San Raffaele University Hospital, Italy (Other); University of Foggia (Other); Azienda Ospedaliera Niguarda Cà Granda (Other); Azienda Policlinico Umberto I (Other); Federico II University of Naples, Department of Clinical Medicine and Surgery, Naples, Italy (Unknown); Città di Lecce Hospital (Unknown); Policlinico G . Martino, Messina Italy (Unknown); Azienda Ospedaliera Universitaria Senese (Other); Azienda Sanitaria di Firenze (Other); Ospedale San Luca, Istituto Auxologico Italiano, Milano (Unknown); Casa di Cura Mater Dei (Unknown); University of Bari (Other); Azienda Ospedaliera di Perugia (Other); I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Italy (Unknown); IRCCS Multimedica (Other); Ospedali Riuniti Ancona (Other); ASST Papa Giovanni XXIII, Bergamo, Italy (Unknown); S. Andrea Hospital (Other); Istituti Clinici Scientifici Maugeri SpA (Other); Istituto Auxologico Italiano - IRCCS - Ospedale San Luca - Milano (Unknown); Azienda Ospedaliero-Universitaria Senese (Unknown); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other); Federico II University (Other); Ospedale Guglielmo da Saliceto, Piacenza (Unknown)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, Professor, Centro Cardiologico Monzino
Other Study IDs: CCM 04-21PA
Record Dates: First submitted 2025-03-10; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
Keywords: prognosis; risk score; heart failure; cardiopulmonary exercise test; exercise
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Heart failure patients: Patients with systolic heart failure, able to exercise

SUMMARY:
Heart failure is a complex condition involving multiple organs beyond the cardiovascular system, all influencing disease progression and prognosis. Accurate risk assessment requires considering multiple variables, as no single parameter alone provides a complete prognostic picture.

This has led to the development of prognostic models combining clinical and laboratory parameters. Some of these models incorporate cardiopulmonary exercise testing (CPET), which provides key prognostic indicators. Since the 1990s, CPET has been recommended in heart failure management guidelines due to its strong prognostic value when combined with clinical data.

However, existing risk models often exclude important predictors such as ventilatory parameters from CPET (VE/VCO₂), renal function, and hemoglobin levels. To address this gap, in 2012 the investigators developed the MECKI (Metabolic Exercise test data combined with Cardiac and Kidney Indexes) score, integrating oxygen consumption, ventilatory efficiency, and easily accessible biochemical and echocardiographic parameters. Unlike previous models requiring extensive data collection, MECKI is based on only six variables, making it practical and effective.

Recent studies suggest the need to update the cutoff values and parameters used for risk stratification, as new therapies and treatment strategies may significantly alter prognostic accuracy in different patient populations.

This study aims to expand and refine the MECKI score by updating the patient dataset, optimizing its performance in specific subgroups, and aligning it with emerging therapeutic approaches.

Additionally, the investigators will evaluate whether the model's risk accuracy varies in advanced-stage patients, those with comorbidities, or under different treatment regimens. This could lead to correction factors that enhance the score's predictive power across diverse clinical scenarios, further improving its applicability and reliability in heart failure management.

DETAILED DESCRIPTION:
Heart failure is a complex condition affecting multiple organs beyond the cardiovascular system, influencing disease progression and prognosis. It has become increasingly evident that accurate risk assessment requires considering multiple variables, as no single parameter alone is sufficient for prognosis.

These findings have led to the identification and study of prognostic parameters that, when combined, allow for a more precise risk estimation and identification of high-risk patients. Various prognostic scores have been developed, utilizing algorithms that integrate multiple variables to estimate an individual's mortality risk. Some scores are based on clinical evaluation and comorbidities, others on laboratory findings, baroreflex sensitivity, heart rate, sleep abnormalities, echocardiographic imaging, or cardiopulmonary exercise testing (CPET), either alone or in combination with other factors.

CPET provides several parameters strongly correlated with prognosis. Since the 1990s, its use-alongside clinical data-has been recommended in heart failure management guidelines. More recently, in addition to peak oxygen consumption, the VE/VCO₂ slope has been recognized as a key prognostic marker, reflecting ventilatory efficiency and ventilation-perfusion mismatch, and has been included in heart transplant assessment criteria.

Current risk models in heart failure often omit important prognostic parameters, such as ventilatory indices from CPET, renal function, and hemoglobin levels. Among the numerous prognostic scores available, only the HF Survival Score (HFSS) and the HF Action Predictive Risk Score Model incorporate exercise-related parameters (peak VO₂ in the former and exercise duration in the latter), yet both neglect ventilatory aspects. Even the widely used Seattle Score does not include exercise-related variables.

In 2012, the researchers developed the MECKI (Metabolic Exercise test data combined with Cardiac and Kidney Indexes) score, integrating oxygen consumption, ventilatory efficiency, and easily accessible biochemical and echocardiographic parameters. Unlike previous models requiring extensive data collection, MECKI is based on just six key variables, making it both practical and effective.

Recent studies indicate the need to review and update the cutoff values and parameters used in prognostic models, as the introduction of new therapies and treatment strategies may significantly impact their predictive power in specific patient populations.

Study Objectives and Purpose The aim of this study is to expand and update the patient dataset to further develop the MECKI score, optimizing its application in patient subgroups and adapting it to new therapies and treatments introduced in clinical practice.

Additionally, the researchers seek to determine whether risk prediction accuracy varies in advanced-stage patients, those with comorbidities, or those receiving different treatments. This could lead to the development of correction factors for the MECKI score, improving its predictive power and applicability across different clinical scenarios.

Study Population Patients with systolic heart failure, consecutively enrolled and followed at multiple Heart Failure Units across Italy.

Patients undergo assessment through medical history collection, physical examination, laboratory tests, ECG, transthoracic echocardiography, and cardiopulmonary exercise testing (CPET).

Follow-up will be conducted according to the protocol of the respective Heart Failure Unit. The follow-up period ends at the last evaluation at the reference center, or upon the patient's death or heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age >18 past or present heart failure (NYHA functional class I-III, stage C of the ACC/AHA classification)
* documentation of left ventricular systolic dysfunction (LVEF <40%)
* stable clinical conditions
* previous or concomitant cardiopulmonary exercise test

Exclusion Criteria:

* scheduled cardiovascular treatment
* clinical unstable condition
* History of pulmonary embolism, significant valvular disease, pericardial disease, severe COPD, exercise-induced angina, exercise-induced ECG changes, severe brady- or tachyarrhythmias, or the presence of comorbidities that interfere with exercise performance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with past or present heart failure (with previous documentation of left ventricular systolic dysfunction (LVEF <40%)), in stable clinical conditions, who underwent a cardiopulmonary exercise test, with no scheduled cardiovascular treatment.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk score | From enrollment to endpoint occurence (death, LVAD implantation, heart transplant) within 15 years
  Expand and update the patient dataset to further develop the Metabolic Exercise test data combined with Cardiac and Kidney Indexes (MECKI) score, optimizing its application in specific patient subgroups and aligning it with newly introduced therapies and treatments in clinical practice.
End point | From enrollment to endpoint occurence (death, LVAD implantation, heart transplant) within 15 years
  Time to Cardiovascular death or LVAD implantation or heart transplant

CONTACTS AND LOCATIONS:
Locations (26):
- Italy (26):
  - Centro Cardiologico Monzino, Milan, Italy
  - Ospedali Riuniti di Ancona, Ancona
  - Istituti Clinici Scientifici Maugeri Bari, Bari
  - Ospedale papa Giovanni XXIII, Bergamo
  - Spedali Civili Brescia, Brescia
  - Spedali Civili, Brescia
  - Università di Foggia, Foggia
  - I.R.C.C.S. Ospedale San Raffaele, Milan
  - IRCCS Istituto Auxologico Italiano, Milan
  - IRCCS Multimedica- Ospedale San Giuseppe, Milan
  - Istituti Clinici Scientifici Maugeri Milano, Milan
  - Ospedale Cà Granda- A.O. Niguarda, Milan
  - Federico II hospital, Naples
  - Azienda Ospedaliera dei Colli - Ospedale Monaldi, Napoli
  - Università degli Studi di Napoli Federico II, Napoli
  - Istituto Mediterraneo per i Trapianti e Terapie ad alta specializzazione, Palermo
  - Ospedale Guglielmo da Saliceto, Piacenza
  - Fondazione Gabriele Monasterio, Pisa
  - Azienda Ospedaliera San Camillo-Forlanini, Roma
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Azienda Ospedaliero-Universitaria Policinico Umberto I, Rome
  - Santo Spirito Hospital, Rome
  - IRCCS Policlinico San Donato, San Donato Milanese
  - S. Maria alle Scotte Hospital UOC cardiologia clinico-chirurgica (UTIC), Siena
  - S. Maria alle Scotte Hospital UOSA malattie cardiovascolari, Siena
  - Azienda sanitaria universitaria Giuliano Isontina (ASUGI), Trieste